CLINICAL TRIAL: NCT04034108
Title: Early Surgical Intervention Combined With Weight-supported Walking Training Improves Neurological and Locomotor Recoveries in 339 Clinically Complete Human Spinal Cord Injuries
Brief Title: Early Surgical Intervention Combined With Weight-supported Walking Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kunming Tongren Hospital (Industry)
Responsible Party: Principal Investigator, Hui Zhu, Director of Department, Kunming Tongren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KunmingTH_HZ_002
Record Dates: First submitted 2019-07-17; First posted 2019-07-26 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Spinal Cord Injuries
Keywords: surgical intervention; decompression; walking training; functional recovery; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiment group (Experimental): All the patients were classified as AIS-A at the time of admission to the clinical center. The MRI was performed in all cases prior to and after the surgery. Surgeries were performed between 12 hours to 30 days after trauma. At 15 days after surgery, with protection of a tailored chest-waist cast made of polyurethane 8 foam for thoracic/lumbar injuries or a neck support for cervical injuries, the patients were encouraged to start weight-supported ambulation training under careful protection by the trainers.
  Interventions: Procedure: Surgical intervention combined with weight-supported ambulation training

INTERVENTIONS:
Procedure: Surgical intervention combined with weight-supported ambulation training — Surgeries were performed between 12 hours to 30 days after trauma. Internal fixation was implemented once instability of the injured spinal column was confirmed by radiology and exploration during operation. At 15 days after surgery, the patients were encouraged to start weight-supported ambulation training under careful protection by the trainers, the patients were encouraged to start weight-supported ambulation training under careful protection by the trainers. The training program was named "Kunming Locomotor Training Program (KLTP)"formulated by actively walking for a duration of 6 hours per day, 6 days per week for a minimum of 6 months.

SUMMARY:
To determine the efficacy of a novel combinatorial treatment involving early surgical intervention and long-term weight-bearing walking training in spinal cord injury (SCI) patients clinically diagnosed as complete or American Spinal Injury Association Impairment Scale Class A (AIS-A).

DETAILED DESCRIPTION:
In the present study, the investigators reported the efficacy of a novel combinatorial approach involving early surgical intervention and long-term weight-bearing walking training in SCI patients clinically defined as complete or AIS-A. The surgical intervention involves the intradural decompression (via durotomy), and, in some cases, intraspinal decompression (via myelotomy). In addition, the investigators had developed a weight-bearing walking training program named "Kunming Locomotion Training Program (KLTP)" to train the patient to walk actively for a duration of 6 hours per day, 6 days per week for a minimum of 6 months (6-6-6 KLTP). The investigators reasoned that early surgical intradural and/or intraspinal decompression would release the intraspinal pressure and, therefore, spare surrounding tissues that would otherwise degenerate during the course of secondary injury. The investigators further reasoned that long-term weight-bearing walking training would "retrain" the residual spinal pathways facilitating recovery of locomotor function, and that a combination of the two would result in even greater functional recoveries.

ELIGIBILITY:
Inclusion Criteria:

* injury levels included cervical, thoracic and lumbar spinal levels;
* neurological examination was AIS-A;
* diagnosis of SCI was confirmed by MRI.

Exclusion Criteria:

* penetrating injuries that caused complete transection of the spinal cord;
* patients with severe brain injuries or other neurological disorders;
* patients with lower motoneuron diseases;
* patients with other conditions including pregnancy, and significant medical, infectious, and psychiatric conditions.

Ages: 4 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2000-05-01 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-05-01 (Actual)

PRIMARY OUTCOMES:
Change of Kunming Locomotor Scale (KLS) | Before surgery, Day 15, Month 3, and Month 6
  Kunming Locomotor Scale is a 10-grade Roman numeral locomotion scoring system. Grade I, the patient can not stand; grade II, the patient is able to stand with weight support and help in fixing the knee; grade III, the patient is able to stand with weight support; grade IV, the patient is able to walk with wheeled weight support and help in fixing the knee of the weight bearing leg; grade V, the patient is able to walk with wheeled weight support; grade VI, the patient is able to walk with the help of a light four-leg support; grade VII, the patient is able to walk with a pair of crutches; grade VIII, the patient is able to walk with a cane; grade IX, the patient is able to walk without support but staggeringly; and grade X, the patient is able to walk stably without support.

SECONDARY OUTCOMES:
Change of American Spinal Injury Association Impairment Scale (AIS) | Before surgery (baseline), Day 15, Month 3, and Month 6
  American Spinal Injury Association Impairment Scale (AIS), as international standards for neurological classification of spinal cord injury, is a 5 point ordinal scale to identify patient's sensory and motor levels, from AIS-A (complete SCI) to AIS-E (normal sensory and motor function).
Magnetic Resonance Imaging | Before surgery
  Magnetic Resonance Imaging (MRI) are performed prior to the surgery to provided important measures determining the injury level, severity, and indication of a surgical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhu, Principal Investigator — Kunming Tongren Hospital
Locations (2):
- China (2):
  - Kunming General Hospital of Chengdu Military Command, Kunming, Yunnan
  - Kunming Tongren Hospital, Kunming, Yunnan

REFERENCES:
- [Derived] Liu Y, Xie JX, Niu F, Xu Z, Tan P, Shen C, Gao H, Liu S, Ma Z, So KF, Wu W, Chen C, Gao S, Xu XM, Zhu H. Surgical intervention combined with weight-bearing walking training improves neurological recoveries in 320 patients with clinically complete spinal cord injury: a prospective self-controlled study. Neural Regen Res. 2021 May;16(5):820-829. doi: 10.4103/1673-5374.297080. PMID 33229715